CLINICAL TRIAL: NCT00226785
Title: A Prospective, Multi-Centre, Randomised, Double-Blind Comparison of Intravenous Dexmedetomidine With Propofol/Midazolam for Continuous Sedation (24 Hours to 14 Days) of Ventilated Patients in Intensive Care Unit
Brief Title: Dexmedetomidine for Continuous Sedation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3005011
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
The study aims to demonstrate that dexmedetomidine is non-inferior to current best practice sedation with propofol/midazolam and daily sedation stops, in maintaining a target depth of sedation in long-stay intensive care unit (ICU) patients, and that dexmedetomidine, compared with current best practice, reduces the length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Clinical need for sedation and mechanical ventilation
* Receiving full intensive care life support
* Expected stay in ICU of at least 48 hours (h) from time of admission
* Expected requirement for sedation of at least 24h from time of randomisation
* Written informed consent within 36h of ICU admission

Exclusion Criteria:

* Acute severe neurological disorder
* Acute uncompensated circulatory failure at time of randomisation
* Severe bradycardia
* Atrioventricular (AV) conduction block (II-III) unless pacemaker fitted
* Severe hepatic impairment
* Need for muscle relaxation at time of randomisation
* Loss of hearing or vision or any condition interfering significantly with RASS assessment
* Positive pregnancy test or currently lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2005-10; Study Completion 2006-07

PRIMARY OUTCOMES:
Proportion of time during sedative infusion with a Richmond Agitation Sedation Scale (RASS) score within the individually-prescribed target range
Time from ICU admission to discharge

SECONDARY OUTCOMES:
Nurse's assessment of subject communication
Duration of mechanical ventilation, weaning time and ventilator-free days in ICU
Length of total hospital stay
Functional recovery during hospitalisation
Need for rescue medication to maintain sedation
Frequency of delirium
Frequency of organ failures and failure-free days
Frequency of critical illness polyneuropathy
ICU- and in-hospital survival
Cost of care in the ICU
Total cost of hospitalisation
Blood levels of dexmedetomidine seen with long-term treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Takala, MD, PhD, Study Chair — University/University Hospital, Bern, Switzerland; Esko Ruokonen, MD, PhD, Principal Investigator — Kuopio University Hospital, Finland; Stephan Jakob, MD, PhD, Principal Investigator — University Hospital, Bern, Switzerland
Locations (4):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Ruokonen E, Parviainen I, Jakob SM, Nunes S, Kaukonen M, Shepherd ST, Sarapohja T, Bratty JR, Takala J; "Dexmedetomidine for Continuous Sedation" Investigators. Dexmedetomidine versus propofol/midazolam for long-term sedation during mechanical ventilation. Intensive Care Med. 2009 Feb;35(2):282-90. doi: 10.1007/s00134-008-1296-0. Epub 2008 Sep 16. PMID 18795253